CLINICAL TRIAL: NCT01775475
Title: Randomized, Phase II Trial of CHOP vs. Oral Chemotherapy With Concomitant Antiretroviral Therapy in Patients With HIV-Associated Lymphoma in Sub-Saharan Africa
Brief Title: Intravenous Chemotherapy or Oral Chemotherapy in Treating Patients With Previously Untreated Stage III-IV HIV-Associated Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC-068; NCI-2012-01695 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U01CA121947 (NIH)
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Results first posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: AIDS-related Diffuse Large Cell Lymphoma; AIDS-related Diffuse Mixed Cell Lymphoma; AIDS-related Diffuse Small Cleaved Cell Lymphoma; AIDS-related Immunoblastic Large Cell Lymphoma; AIDS-related Lymphoblastic Lymphoma; AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Small Noncleaved Cell Lymphoma; Stage III AIDS-related Lymphoma; Stage IV AIDS-related Lymphoma
MeSH Terms: conditions — Lymphoma, AIDS-Related | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Lomustine; Etoposide; Procarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (CHOP) (Active Comparator): Patients receive CHOP chemotherapy comprising cyclophosphamide IV on day 1, doxorubicin hydrochloride IV on day 1, vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Drug: prednisone; Other: laboratory biomarker analysis
- Arm II (oral chemotherapy) (Experimental): Patients receive lomustine PO QD on day 1 (courses 1 and 3 only), etoposide PO QD on days 1-3, cyclophosphamide PO QD on days 22-26, and procarbazine hydrochloride PO QD on days 22-26. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lomustine; Drug: etoposide; Drug: cyclophosphamide; Drug: procarbazine hydrochloride; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
  Arms: Arm I (CHOP)
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
  Arms: Arm I (CHOP)
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
  Arms: Arm I (CHOP)
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra
  Arms: Arm I (CHOP)
Drug: lomustine — Given PO
  Other Names: Belustine; CCNU; CeeNU
  Arms: Arm II (oral chemotherapy)
Drug: etoposide — Given PO
  Other Names: EPEG; VP-16; VP-16-213
  Arms: Arm II (oral chemotherapy)
Drug: cyclophosphamide — Given PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
  Arms: Arm II (oral chemotherapy)
Drug: procarbazine hydrochloride — Given PO
  Other Names: Ibenzmethyzin; Matulane; MIH; Natulan; PCB
  Arms: Arm II (oral chemotherapy)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well intravenous (IV) chemotherapy or oral chemotherapy works in treating patients with previously untreated stage III-IV human immunodeficiency virus (HIV)-associated non-Hodgkin lymphoma. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, prednisone, lomustine, etoposide, and procarbazine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the efficacy of standard cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone (CHOP) and an oral chemotherapy regimen for acquired immune deficiency syndrome (AIDS)-related (AR)-non-Hodgkin lymphoma (NHL) in sub-Saharan Africa with respect to overall survival (OS).

SECONDARY OBJECTIVES:

I. To compare the objectives response rate (ORR) of persons randomized to CHOP and oral chemotherapy.

II. To compare the progression free survival (PFS) of persons randomized to CHOP and oral chemotherapy.

III. To compare the safety and tolerance of persons randomized to CHOP and oral chemotherapy.

TERTIARY OBJECTIVES:

I. To describe the rates of completion of therapy of persons randomized to CHOP and oral chemotherapy.

II. To describe adherence to chemotherapy of persons randomized to CHOP and oral chemotherapy.

III. To describe adherence to antiretroviral therapy of persons randomized to CHOP and oral chemotherapy.

IV. To describe the effects of therapy on HIV control, as measured by cluster of differentiation (CD)4 counts and HIV viral load.

V. To investigate correlates of survival.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive CHOP chemotherapy comprising cyclophosphamide intravenously (IV) on day 1, doxorubicin hydrochloride IV on day 1, vincristine sulfate IV on day 1, and prednisone orally (PO) on days 1-5. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive lomustine PO once daily (QD) on day 1 (courses 1 and 3 only), etoposide PO QD on days 1-3, cyclophosphamide PO QD on days 22-26, and procarbazine hydrochloride PO QD on days 22-26. Treatment repeats every 6 weeks for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to provide written informed consent to participate
* Adults, 18 years of age or older; date of birth should be determined based on the best possible information or source documentation available
* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or confirmed by HIV-1 antigen or plasma HIV-1 ribonucleic acid (RNA) viral load > 1,000 copies/mL

  * NOTE: the term "licensed" refers to a United States (U.S.) Food and Drug Administration (FDA)-approved kit or for sites located in countries other than the United States, a kit that has been certified or licensed by an oversight body within that country and validated internally
  * WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment; a reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load
* Biopsy-proven, measurable or assessable systemic NHL that has been confirmed by an AIDS Malignancy Clinical Trial Consortium (AMC)-approved site pathologist; if a hard copy of the pathology report is unavailable at the time of enrollment, a verbal report by the pathologist confirming the diagnosis must be documented in the medical chart
* Pathology slides from tumor tissue obtained by surgical excision or core biopsy must be reviewed by the designated site pathologist, or backup pathologist, prior to study entry; confirmation of the diagnosis must be documented by the AMC-approved pathologist prior to study entry; please reference the AMC-068 Manual of Procedures (MOP) for further instructions on documenting the diagnosis; the site pathologist for NHL must be approved through the AMC's external quality assessment (EQA) process
* Participants must have fifteen blank(unstained) slides or a diagnostic tissue block must be available for central pathology review by the AMC Core Pathology Laboratory
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Participants must have an estimated life expectancy of > 6 weeks
* White blood cells (WBC) >= 3,000 cells/uL (3.0 x 10^9 L) or
* Absolute granulocytes >= 1500 cells/uL (1.5 x 10^9 L)
* Platelets >= 100,000 cells/uL (75 x 10^9 L)
* Hemoglobin > 8 g/dL (5.0 mmol/L)
* Patients may enroll with lower hematologic values, if bone marrow involvement is documented; in this case, patients should be transfused to hemoglobin > 8 g/dL
* Serum creatinine < 3.0 mg/dL (265.2 umol/L)
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN), unless elevated secondary to lymphomatous involvement of liver or biliary system, or due to other HIV medications (e.g., indinavir, tenofovir, or atazanavir); if secondary to lymphomatous involvement, an initial upper limit of total bilirubin 5 mg/dL (85.5 uM/L) should be utilized - for direct bilirubin > 1.2 mg/dL (20.5 uM/L)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 institutional ULN (unless elevated secondary to lymphomatous involvement of the liver)
* Participants must have a lumbar puncture with negative cerebral spinal fluid cytology within 6 weeks prior to enrollment; participants must be without evidence for central nervous system (CNS) lymphoma on neurological exam and have no radiographic evidence (if radiographic studies are done) of CNS lymphoma (inclusive of parenchymal, vitreal, or leptomeningeal involvement)
* Participants must not have had any prior chemotherapy or radiation therapy and no more than 10 days of corticosteroids in the preceding 30 days prior to enrollment
* All participants must be prescribed combination antiretroviral therapy with the goal of virological suppression using an acceptable regimen that adheres to national guidelines for treatment of HIV infection; non-suppressed, treatment experienced patients, defined as patients with a viral load > 400 copies/mL who have been on antiretroviral therapy for more than 4 months can be enrolled if an alternative antiretroviral therapy (ART) regimen is available that includes at least two ART drugs that, in the opinion of the site investigator, are expected to have activity based on genotypic testing (if available) and treatment history; patients are not allowed to receive zidovudine (azidothymidine [AZT]) as part of concurrent chemotherapy and ART regimen, since it is myelosuppressive; zidovudine may be discontinued and substituted as clinically indicated prior to or at the time of enrollment.
* Participants of childbearing potential, defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months), must have a pregnancy test within 7 days prior to enrollment and agree to use an effective form of contraception (e.g., barrier contraception, highly effective hormonal contraception)
* Participants are allowed to have an active infection(s) for which they are receiving drug treatment provided the clinical status is judged to be stable and survival is estimated to be at least 6 weeks
* Participants must, in the opinion of the investigatory, be capable of complying with the protocol
* Participants must be able to take oral medications
* Participants must have a CD4 count performed within 30 days of enrollment

Exclusion Criteria:

* Inability to provide informed consent
* A medical or psychiatric illness that precludes ability to give informed consent or is likely to interfere with the ability to comply with the protocol stipulations
* Participants with circumstances that will not permit completion of the study or required follow-up; for instance, if travel to and from treatment site is an issue
* Pregnant or breastfeeding
* Inability to swallow oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Strother, Principal Investigator — AIDS Associated Malignancies Clinical Trials Consortium
Locations (2):
- Moi Teaching and Referral Hospital, Eldoret, Kenya
- University of Zimbabwe College of Health Sciences, Harare, Zimbabwe

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (CHOP) | Arm II (Oral Chemotherapy)
Started | 4 | 3
Completed | 1 | 0
Not Completed | 3 | 3
Not completed — Death | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (CHOP) | Arm II (Oral Chemotherapy) | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Median (Full Range); unit: years] | 52.5 [43.0 to 55.0] | 46.0 [39.0 to 47.0] | 47.0 [39.0 to 55.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Zimbabwe | 1 | 0 | 1
  Kenya | 1 | 2 | 3
  Malawi | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Proportion of participants who survived 2 years
Time Frame: Up to 24 months
Population: Study participants whose survival status was known at two years.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm I (CHOP) | Arm II (Oral Chemotherapy)
Number analyzed (Participants) | 3 | 3
Proportion of participants | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: Overall Response Rate
Description: Overall response is complete or partial response as defined by response definitions of the 2014 International Conference on Malignant Lymphoma Imaging Working Group (i.e. Lugano classification). Complete response is the disappearance of all lesions with no new lesions detected. Partial response is >=50% decrease in the sum of the perpendicular diameters of up to 6 target measurable nodes and extranodal sites and no new sites of disease.
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (CHOP) | Arm II (Oral Chemotherapy)
Number analyzed (Participants) | 4 | 3
Participants | 3 | 1

3. Primary Outcome: Progression-free Survival
Description: Proportion of participants who survived without disease progression at 2 years
Time Frame: Up to 24 months
Population: Participants whose disease and survival status were known at 2 years
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Arm I (CHOP) | Arm II (Oral Chemotherapy)
Number analyzed (Participants) | 3 | 3
proportion | 0 [0 to 0] | 0 [0 to 0]

4. Primary Outcome: Participants Who Experienced an Adverse Event
Description: Number of participants who experienced an adverse event
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (CHOP) | Arm II (Oral Chemotherapy)
Number analyzed (Participants) | 4 | 3
Participants | 4 | 3

5. Primary Outcome: Number of Patients Who Complete Treatment
Description: Number of patients who complete chemotherapy treatment.
Time Frame: Up to 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (CHOP) | Arm II (Oral Chemotherapy)
Number analyzed (Participants) | 4 | 3
Participants | 3 | 1

6. Primary Outcome: Proportion of Patients Who Are Adherent to Antiretroviral Therapy
Description: Number of patients who did not miss any of their doses of antiretroviral therapy
Time Frame: Up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (CHOP) | Arm II (Oral Chemotherapy)
Number analyzed (Participants) | 4 | 3
Participants | 3 | 3

7. Primary Outcome: Proportion of Patients Who Are Adherent to Chemotherapy
Description: Patients who did not miss any doses of chemotherapy
Time Frame: Up to 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (CHOP) | Arm II (Oral Chemotherapy)
Number analyzed (Participants) | 4 | 3
Participants | 4 | 3

8. Primary Outcome: Change in Absolute CD4 Count From Baseline to Post-treatment
Description: Change in absolute CD4 count from baseline to post-treatment (visit 6)
Time Frame: From baseline to 18 weeks
Population: Participants who had absolute CD4 count measurements at baseline and visit 6
Measure: Mean (Standard Deviation); unit: cells per mm^3
Arm/Group | Arm I (CHOP) | Arm II (Oral Chemotherapy)
Number analyzed (Participants) | 3 | 3
cells per mm^3 | -41.3 (136.5) | 203.3 (153.1)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Arm I (CHOP) | Arm II (Oral Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 3/4 | 3/3
Serious Adverse Events (participants affected / at risk) | 4/4 | 3/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (CHOP) (N=4) | Arm II (Oral Chemotherapy) (N=3)
Neoplasms, other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Fatigue (General disorders) | 1 | 0
Encephalitis infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Fever (General disorders) | 0 | 1
Death cause unknown (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (CHOP) (N=4) | Arm II (Oral Chemotherapy) (N=3)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Blood and lymphatic system disorders, other (Blood and lymphatic system disorders) | 1 | 1
Tinnitus (Eye disorders) | 0 | 1
Blurred vision (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Alkaline phosphatase (Investigations) | 1 | 2
GGT increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 1
White blood cell decreased (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Facial nerve disorder (Nervous system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Nail coloration (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT01775475/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT01775475/ICF_001.pdf